CLINICAL TRIAL: NCT02762786
Title: Effectiveness of Musical Training in the Improvement of Psychological Well-being and Quality of Life of Children From Low Income Families
Brief Title: Effectiveness of Musical Training in Children From Low Income Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PhD_2
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Child

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Participants in the experimental group will receive weekly one-hour lessons on musical training for 12 weeks, conducted by the Music Children Foundation. The Music Children Foundation is a non-governmental organization established by a group of professional musicians with the objective of transforming children's lives and instils positive values in the entire community through music. It aims to provide free musical training to low-income children and children with chronic diseases, including those with Down's syndrome, mucopolysaccharidoses, skeletal dysplasia and visual impairment.
  Interventions: Behavioral: musical training
- Wait-list control group (No Intervention): Participants in the waitlist control group will receive the same training after the experimental group had completed the intervention.

INTERVENTIONS:
Behavioral: musical training — The subjects in the experimental group will receive weekly one-hour lessons on musical training for 12 weeks, conducted by the Music Children Foundation.
  Arms: Experimental

SUMMARY:
This study aims to examine the effectiveness of musical training in promoting happiness and quality of life of preschool children from low-income families.

Participants in the experimental group will attend a weekly 1-hour musical training lesson for 12 weeks conducted by the Music Children Foundation. While participants in the waitlist control group received the same training after the experimental group had completed the intervention.

DETAILED DESCRIPTION:
Children from low income families generally suffer from hard conditions,such as poor living conditions, inadequate nutrition, and delay in accessing health care services. Such problems may made children suffer from developmental problems and malnutrition and to have a lower level of intelligence and difficulties in language comprehension, which may not only have profound impacts on children's physical well-being, but on their psychological well-being as well. Musical training is considered to have potential for promoting psychological well-being among children mostly because music is found to be important to a child's early psychological development. A growing number of educators and researchers suggest that, of all the stages of life, infancy may be the time when music has the most important impact on an individual. Babies hear language long before they are able to comprehend it. The quality and the quantity of what is unconsciously absorbed in infancy relates directly to later development. Musical training has been used for various purposes such as improving language development, self-expression, memory skills, concentration, social interaction, fine motor skills, listening, problem-solving, teamwork, goal setting, and coordination. More importantly, when a child learns to sing and play music, other areas of development - creativity, family bonding, self-esteem, confidence, emotional development - are also positively impacted.

Nevertheless, although musical training is popular and is considered to be a beneficial intervention in the promotion of psychological well-being, longitudinal studies that examine the efficacy of music-making in children from low-income families are limited. Importantly, there is to date no study that examines the effects of musical training on enhancing the psychological well-being among these children. There is an imperative need for rigorous empirical scrutiny of the effectiveness of musical training in promoting the psychological well-being of children from low-income families. Therefore, the aim of this study is to examine the effectiveness of musical training in promoting happiness and quality of life of preschool children from low-income families.

ELIGIBILITY:
Inclusion Criteria:

* be aged from 3 to 6 years,
* be able to communicate in Cantonese,
* be from low-income families; that is, less than half the median monthly household income or recipients of Comprehensive Social Security Assistance.

Exclusion Criteria:

* children who had studied or were studying (at the time of the intervention) a musical instrument
* children who were receiving other community services at the time of the intervention,
* children with chronic illness or identified cognitive and learning problems.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 171 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
The change of quality of life from baseline at 12 weeks follow-up between intervention and control group. | 12 weeks follow-up
  The subjects' quality of life will be assessed at 12 weeks after starting the intervention, using the Chinese version of the Paediatric Quality of Life Inventory 4.0 Generic Core Scale (PedsQL 4.0).
  The parents will be asked to fill in this questionnaire for their children. The PedsQL is designed to measure children's healthrelated quality of life. It comprises 23 items rated on a 5-point Likert scale. These items are categorised into four domains: physical functioning (eight items), emotional functioning (five items), social functioning (five items) and school functioning (five items). The total possible range of scores is from 0 to 100, with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Quality of life at baseline between intervention and control group. | baseline
  The subjects' quality of life will be assessed at the baseline, using the Chinese version of the Paediatric Quality of Life Inventory 4.0 Generic Core Scale (PedsQL 4.0) The parents will be asked to fill in this questionnaire for their children. The PedsQL is designed to measure children's healthrelated quality of life. It comprises 23 items rated on a 5-point Likert scale. These items are categorised into four domains: physical functioning (eight items), emotional functioning (five items), social functioning (five items) and school functioning (five items). The total possible range of scores is from 0 to 100, with higher scores indicating better quality of life.
Happiness at baseline between intervention and control group. | baseline
  The subjects' happiness will be assessed 12 weeks after starting the intervention, using the Visual Analog Scale.
  The children will be asked to rate their average level of happiness in the last week from zero (not happy or sad) to ten (extremely happy), with higher scores representing higher level of happiness.
The change of happiness from baseline at 12 weeks follow-up between intervention and control group. | 12 weeks follow-up
  The subjects' happiness will be assessed 12 weeks after starting the intervention, using the Visual Analog Scale.
  The children will be asked to rate their average level of happiness in the last week from zero (not happy or sad) to ten (extremely happy), with higher scores representing higher level of happiness.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ho LLK, Li WHC, Cheung AT, Xia W, Ho KY, Chung JOK. Low-income parents' perceptions of the importance of a musical training programme for their children: a qualitative study. BMC Public Health. 2020 Sep 25;20(1):1454. doi: 10.1186/s12889-020-09568-7. PMID 32977785